CLINICAL TRIAL: NCT02123433
Title: Serological Response to Antipneumococcal Vaccination and Consequent Impact on Streptococcus Pneumoniae Nasal Carriage in HIV Positive Adults: a Prospective Study Using 13-valent Conjugate Vaccine
Brief Title: Serological Response to Antipneumococcal Vaccination and Impact on Streptococcus Pneumoniae Nasal Carriage in HIV Adults
Acronym: PCV13HIV2011
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Siena (Other)
Collaborators: Ministry of Education, Universities and Research, Italy (Other)
Responsible Party: Principal Investigator, Francesca Montagnani, Assistant Professor, University of Siena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-004518-40; 2011-004518-40 (EudraCT Number)
Record Dates: First submitted 2013-12-13; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infection; Pneumococcal Infections
Keywords: HIV; Streptococcus pneumoniae; 13-valent conjugate pneumococcal vaccine; Vaccine; Immunological Response; Pneumococcal Carriage
MeSH Terms: conditions — HIV Infections; Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

ARMS (1):
- 13-valent vaccine (Experimental)
  Interventions: Biological: pneumococcal conjugate 13 valent vaccine

INTERVENTIONS:
Biological: pneumococcal conjugate 13 valent vaccine — Pneumococcal polysaccharide conjugate vaccine(13-valent adsorbed) conjugated to CRM197 carrier protein and adsorbed on aluminum phosphate (0.125 mg of aluminum).
  Pharmaceutical form: suspension for injection. Dosage: 0.5 ml, containing 2.2 g of polysaccharide for serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F, and 4.4 micrograms for serotype 6B.
  Prevenar 13 is administered in two doses,each of 0.5 ml, with an interval of 2 months, injected intramuscularly in the deltoid muscle of the arm.
  Other Names: Prevenar13

SUMMARY:
S. pneumoniae is frequently isolated from nasal swabs of healthy subjects, but it can also cause severe diseases (pneumonia, bacteraemia, meningitis and sepsis).HIV-infected subjects are more sensitive to invasive diseases and recurrent infection than the general population. Nasal carriage is the main pathogenetic feature for invasive disease: bacteraemia is more frequent in carriers, HIV+ patients are constantly colonized by the same pneumococcal strain and their nasopharyngeal isolates have features similar to subsequent invasive strains. A 23-valent polysaccharide vaccine (PPV23) has long been available and recommended in the HIV+ population as prophylaxis for invasive disease. Studies regarding efficacy of PPV23 in HIV+ are controversial and highlight that immune response induced by PPV23 in HIV+ is poor and an hyporesponsiveness to repeated polysaccaridic antigens stimulation can occur. Moreover, PPV23 seems not to affect pneumococcal carriage status and could lead to emergence of non-vaccine serotypes. The conjugation of pneumococcal capsular polysaccharides to carrier proteins results in an improved T-cell dependent immune response, characterized by increased antibody concentrations and induction of T and B memory cells, with a demonstrated higher efficacy in children. A heptavalent vaccine conjugated with diphtheria toxoid (PCV7) is approved in Europe since 2001 and is effective in reducing incidence of invasive disease by vaccine serotypes (4, 6B, 9V, 14, 18C, 19F, 23F), in both children and adults, due to effect of herd immunity. A PCV13 formulation has recently been developed, covering PCV7 serotypes plus 1, 3, 5, 6A, 7F and 19A. PCV13 revealed the same safety profile as PCV7 in pediatric patients, that are the main target of conjugate vaccines licensure. Some trials showed a better antibody response in terms of quantity and quality in HIV + adults by using PCV7 as compared to PPV23. However these data were not unequivocally confirmed in further studies on the use of PCV7 alone or in combination with PPV23. The first trials of PCV13 use in adults showed the same or even better response compared to PPV23, with a safety and tolerability similar to PCV7. PCV13 in HIV+ adults is a promising candidate prophylactic measure for pneumococcal infections. The purpose of this study is to evaluate serological response and prevalence of nasopharyngeal colonization by S. pneumoniae in HIV+ non-hospitalized adults, following vaccination with 2 doses of PCV13.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* obtained informed consent
* outpatient
* CD4 ≥200 cells/µl in the last two evaluations before T0

Exclusion Criteria:

* > 65 years old
* presence of acute infectious disease
* antibiotic therapy (ongoing or in the previous <= 7 days)
* previous PPV23 or PCV7 vaccination
* Pregnancy
* Current immunomodulatory therapy
* Immunosuppression not HIV related

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Serological response after 2 doses of PCV13 vaccine. | Twenty months
  Measure of serological response after 2 doses of PCV13 vaccine (booster dose after 8 weeks) in HIV+ adults.
Pneumococcal nasopharyngeal colonization | Twenty months
  to determine the rate of nasopharyngeal colonization by different pneumococcal serotypes in HIV-positive adults, in relation to baseline antibody titers at T0

SECONDARY OUTCOMES:
Pneumococcal chemosusceptibility | Twenty months
  Number and percentages of antibiotic resistant (including multiresistant) strains
Molecular epidemiology | Twenty months
  Molecular typing combining PFGE (Pulsed Field Gel Electrophoresis), MLST (MultiLocus Sequence Typing) and PCR analysis of bacterial isolates.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Montagnani, MD, PhD, Principal Investigator — Università di Siena
Locations (2):
- Italy (2):
  - Istituto di Clinica delle Malattie Infettive, Policlinico Gemelli, Roma
  - UOC Malattie Infettive Universitarie, Policlinico Le Scotte, Siena

REFERENCES:
- [Derived] Belmonti S, Rossetti B, Modica S, Paglicci L, Borghetti A, Ciccullo A, Picarelli C, Cauda R, De Luca A, Montagnani F, Lombardi F. Long-Term Serological Response to 13-Valent Pneumococcal Conjugate Vaccine Versus 23-Valent Polysaccharide Vaccine in HIV-Infected Adults. Infect Dis Ther. 2019 Sep;8(3):453-462. doi: 10.1007/s40121-019-0256-z. Epub 2019 Jul 30. PMID 31364010
- [Derived] Lombardi F, Belmonti S, Fabbiani M, Morandi M, Rossetti B, Tordini G, Cauda R, De Luca A, Di Giambenedetto S, Montagnani F. Immunogenicity and Safety of the 13-Valent Pneumococcal Conjugate Vaccine versus the 23-Valent Polysaccharide Vaccine in Unvaccinated HIV-Infected Adults: A Pilot, Prospective Controlled Study. PLoS One. 2016 Jun 3;11(6):e0156523. doi: 10.1371/journal.pone.0156523. eCollection 2016. PMID 27258647
- [Derived] Belmonti S, Lombardi F, Morandi M, Fabbiani M, Tordini G, Cauda R, De Luca A, Di Giambenedetto S, Montagnani F. Evaluation and Optimization of an ELISA Procedure to Quantify Antibodies Against Pneumococcal Polysaccharides Included in the 13-Valent Conjugate Vaccine. J Immunoassay Immunochem. 2016;37(2):189-200. doi: 10.1080/15321819.2015.1106949. PMID 26506438